CLINICAL TRIAL: NCT06900712
Title: A Novel, Single-Session Intervention for Sexual Assault-Related Psychopathology Among College Students
Brief Title: Positive Processes and Transition to Health - Single-Session (PATH-SS)
Acronym: PATH-SS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Norah Feeny, Principal Investigator, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20240516
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: PTSD; Depression
Keywords: ptsd; trauma; depression; stressor; posttraumatic stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PATH-SS (Experimental): This single-session intervention includes the following components:
  * Providing the PATH-SS rationale.
  * A review of life events (PATH of life: negative and positive).
  * A verbal narrative of the sexual assault (revisiting and processing as is done in imaginal exposure)
  * Reminiscence and processing of a major positive life event, and real-life practice to enact what was taught. In positive reminiscence, clients vividly remember the positive event providing details and focus on positive emotions. The therapist will encourage savoring of the experience and encourage facial expression of the positive emotions, so that clients do not dampen, avoid, or minimize the experience. This is particularly relevant with depression.
  * Summary of content, integration and consolidation of learning, application of new learning and resilience in real life as next steps.
  Interventions: Behavioral: PATH-SS

INTERVENTIONS:
Behavioral: PATH-SS — This single-session intervention includes the following components:
  * Providing the PATH-SS rationale.
  * A review of life events (PATH of life: negative and positive).
  * A verbal narrative of the sexual assault (revisiting and processing as is done in imaginal exposure)
  * Reminiscence and processing of a major positive life event, and real-life practice to enact what was taught. In positive reminiscence, clients vividly remember the positive event providing details and focus on positive emotions. The therapist will encourage savoring of the experience and encourage facial expression of the positive emotions, so that clients do not dampen, avoid, or minimize the experience. This is particularly relevant with depression.
  * Summary of content, integration and consolidation of learning, application of new learning and resilience in real life as next steps.

SUMMARY:
The goal of this clinical trial is to test a brief, new psychotherapy (called Positive Processes and Transition to Health - Single Session, or PATH-SS) that aims to provide relief for people who are suffering after experiencing a sexual assault. This research will explore whether this new psychotherapy reduces sexual assault related distress, including posttraumatic stress and depression symptoms. The main questions it aims to answer are:

Does PATH-SS leads to improvements in PTSD and depression symptoms (pre- to post- and 1-month follow-up)? Do participants perceive PATH-SS to be acceptable, helpful, and do they complete/adhere to treatment? Participants will complete a pre-treatment/baseline assessment to confirm eligibility, and those who are eligible will receive the single-session intervention and will complete a post-treatment and a 1-month follow-up assessment of stressor-related symptoms.

DETAILED DESCRIPTION:
This study will be an open trial to determine if PATH-SS reduces stressor-related symptoms of PTSD and/or depression after sexual assault in a sample of 45 college students who have experienced a sexual assault. Potential participants will first undergo a pre-screening to assess for likelihood of elegibility. Participants who may be eligible will proceed to the pre-treatment/baseline assessment; those excluded will be given referrals.

After informed consent is obtained, participants will complete the pre-treatment/baseline assessment to confirm eligibility. The assessing clinician will consult with the PI before making eligibility decisions. Eligible participants will then receive one session of the PATH-SS intervention, lasting up to 2 hours.

Symptoms will be assessed pre-treatment, post-treatment, and at 1-month follow-up, with each assessment lasting approximately 1 hour. Participants will be compensated $20 via Amazon gift card for each assessment completed following treatment. Participants will not be compensated for the intervention session.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: from 18 to 65.
2. Has experienced unwanted sexual contact or sexual assault during their time as a college student, with a minimum of 12 weeks since the event and a maximum of 5 years since the event.
3. Enrolled in any undergraduate, graduate, or professional program at a college or university in the state of Ohio.
4. Elevated symptoms on either the Posttraumatic Diagnostic Scale (PDS-5) or the Quick Inventory of Depressive Symptomatology (QIDS-SR), at least moderate: 18 on PDS-5 (Foa et al., 2016) and/or 11 on QIDS (moderate depression severity; Rush et al., 2003), with symptoms persisting for 1 month or longer.

Exclusion Criteria:

1. Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by DSM-5.
2. Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
3. Severe self-injurious behavior or suicide attempt within the previous three months.
4. Currently engaged in cognitive behavioral psychotherapy.
5. No clear memory of the event.
6. Unstable dose of psychotropic medications in prior 3 months.
7. Ongoing intimate relationship with the perpetrator.
8. Current diagnosis of a substance use disorder (DSM-5).
9. Residence outside the state of Ohio.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Scale-Interview (PSS-I-5; Foa et al., 2016) | From baseline to follow-up at 1 month after treatment completion
  The PSS-I is a 24-item, state-of-the-art, psychometrically-validated interview used to assess DSM-5 criteria for PTSD and symptom severity. The PSS-I-5 includes 20 questions assessing symptom severity on a 5-point Likert scale (0 = not at all, 4 = six or more times a week/severe), and scores are calculated by summing responses, with higher scores indicating higher PTSD severity, as well as two questions assessing distress and interference and two questions assessing symptom onset and duration.
Quick Inventory of Depressive Symptomatology-Clinican Report (QIDS-C; Rush et al., 2003) | From baseline to follow-up at 1 month after treatment completion
  The QIDS-C is a 16 item, state-of-the-art, psychometrically-validated interview used to assess depression. Items are rated on a 4-point scale with anchors that vary with the question (e.g., 0 = I do not feel sad, 3 = I feel sad nearly all of the time).
Post-traumatic Stress Diagnostic Scale (PDS-5; Foa et al., 2016) | From baseline to follow-up at 1 month after treatment completion
  The PDS-5 is a 24-item self-report measure used to assess prior trauma exposure and subsequent PTSD symptoms in the past month. The PDS-5 uses a trauma screen to identify prior exposure to traumatic events and assesses the severity of DSM-5 PTSD symptoms related to the event causing the most distress. The PDS-5 includes 20 questions assessing symptom severity on a 5-point Likert scale (0 = not at all, 4 = six or more times a week/severe), and scores are calculated by summing responses, with higher scores indicating higher PTSD severity. The PDS-5 also includes two questions assessing distress and interference and two questions assessing symptom onset and duration.
Quick Inventory of Depressive Symptomatology Self-Report Version (QIDS-SR; Rush et al., 2003) | From baseline to follow-up at 1 month after treatment completion
  The QIDS-SR is a 16-item self-report measure that assesses depression. Items are rated on a 4-point scale with anchors that vary with the question (e.g., 0 = I do not feel sad, 3 = I feel sad nearly all of the time).

SECONDARY OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS; Snaith et al., 1995) | From baseline to follow-up at 1 month after treatment completion
  The SHAPS is a 14-item self-report measuring the capacity to experience pleasure. On a four-point scale (1 = Strongly Agree to 4 = Strongly Disagree), varying statements are rated (e.g., "I would find pleasure in small things"; "I would find pleasure in a telephone call from a friend"). The measure has good convergent and discriminant validity and reflects a unidimensional construct of anhedonia (Leventhal et al., 2006; Nakonezny et al., 2010).
Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988) | From baseline to follow-up at 1 month after treatment completion
  The MSPSS is a 12-item self-report measure that assesses an individual's perceived level of social support from family, friends, and significant others. Items are rated on 7-point Likert scale (1 = Very Strongly Disagree, 7 = Very Strongly Agree).
Working Alliance Inventory - Short Revised (WAI-SR; Munder et al., 2010) | Post-treatment assessment and follow-up at 1 month after treatment completion
  The WAI-SR is a refined measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. The WAI-SR demonstrated good psychometric properties in an initial validation in psychotherapy outpatients in the USA (Munder et al., 2010), as well as in subsequent studies with college students (e.g., Jeong et al., 2023).
Relative Distress and Cost-Benefit Questions (Cromer et al., 2006; DePrince & Freyd, 2004) | Post-treatment assessment and follow-up at 1 month after treatment completion
  Includes three questions measuring participants' experiences of relative distress and cost-benefit beliefs about the survey content: "Was completing study tasks related to the topic of unwanted sexual encounters more or less distressing than anticipated?"; "How important do you believe it is for psychologists to ask about unwanted sexual encounters in order to study the impact of them?"; and "Please consider both your experience completing study tasks related to the topic of unwanted sexual encounters, and your feelings about how important it is that we ask these questions. How good of an idea is it to include such tasks in psychology research?". Items are rated on a 5-point scale with anchors that vary with the question (e.g., 1 = much more distressing, 2 = somewhat more, 3= neutral, 4= somewhat less, and 5 = much less distressing).
Client Satisfaction Questionnaire (CSQ-8; Attkisson & Greenfield, 1994; 2004) | Post-treatment assessment and follow-up at 1 month after treatment completion
  The CSQ-8 is an 8-item questionnaire used to assess satisfaction in mental health services (Sitzia, 1999). This tool includes a brief standardized scale with good psychometric properties that provides an overall assessment of satisfaction (Rush et al. 2008). An additional item was added to specifically assess single-session format of treatment.
Treatment Credibility Scale (CS, Addis & Carpenter, 1999) | Post-treatment assessment and follow-up at 1 month after treatment completion
  The CS is a 6-item self-report questionnaire that was developed for the purpose of the present study to assess patients' perceptions of the credibility of the treatment they were being provided. Participants responded to each item by rat- ing the extent to which the treatment makes sense and is logical to them on a 5-point Likert-type scale ranging from 1 to 5. The six treatment credibility items are: (a) How credible do you think this therapy is? ("not at all credible" to "very credible"); (b) How logical does this therapy seem to you? ("not at all logical" to "very logical"); (c) How much do you trust this therapy to help you? ("not at all" to "very much"); (d) How credible does your therapist seem? ("not at all credible" to "very credible"); (e) How much do you trust your therapist to be able to help you? ("not at all" to "very much"); and (f) How knowledgeable does your therapist appear? ("not at all knowledgeable" to "very knowledgeable").
Utility of Techniques Inventory (UTI; adapted from Foa et al., 2002; Bluett et al., 2014) | Post-treatment assessment and follow-up at 1 month after treatment completion
  This measure consists of 8 items assessing adherence to and utility of skills/techniques taught in therapy. Items are rated on a 5-point Likert scale with anchors that vary with the question (e.g., 0 = Not at all, 4 = More than 10 times; 0 = Not at all helpful, 4 = Extremely helpful).

OTHER OUTCOMES:
Demographics Questionnaire | Baseline
  The demographics questionnaire asks participants to provide information related to their age, sex and gender identity, sexual orientation, ethnicity, relationship status, college year, and living situation (e.g. dormitory, sorority, off-campus).
Treatment History Questionnaire (THQ) | Baseline
  This 4-item measure asks about current and past engagement in mental health services, respectively.
Mini-International Neuropsychiatric Interview (MINI; Sheehan et al., 1998) | Baseline
  The MINI is a brief, structured diagnostic interview used to screen for the major psychiatric disorders according to current diagnostic standards (e.g., the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-5]). Validation and reliability studies have been done comparing the MINI to the structured interviews developed by the American Psychiatric Assocaition and the World Health Organization (e.g., Amorim, 2000; Shields et al., 2021). The results of these studies show that the MINI has similarly high reliability and validity properties to both these instruments, but can be administered in a much shorter period of time (median administration time = 15 minutes).
Columbia-Suicide Severity Rating Scale (C-SSRS; Posner et al., 2008) | From baseline to follow-up at 1 month after treatment completion
  The C-SSRS will be administered by members of the study team (under the supervision of a licensed therapist) used to assess inclusion/exclusion criteria and monitor suicidality.

CONTACTS AND LOCATIONS:
Overall Officials: Norah C Feeny, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No